CLINICAL TRIAL: NCT03138265
Title: Improvements in Aerobic Performance Following a Four-week Period of High Intensity Interval Training in the Elderly.
Brief Title: HIT Training in the Frail Elderly.
Acronym: eHIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: eHIT_Protocol
Record Dates: First submitted 2015-09-21; First posted 2017-05-03 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Sarcopenia; Aged; Exercise; Preoperative Care
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — High-Intensity Interval Training

ARMS (1):
- High intensity exercise training (Experimental): HIT training protocol.
  Interventions: Behavioral: HIIT Device: ergometer

INTERVENTIONS:
Behavioral: HIIT Device: ergometer — Supervised exercise training.
  Other Names: High intensity interval training

SUMMARY:
This pilot study aims to investigate whether high intensity interval training can result in rapid improvements in physical fitness amongst the frail elderly (over 70 years old). Participants will undergo a wide range of physical fitness measures followed by a four week exercise protocol. Determination of improvement will be by repeated testing of the physical measures taken for baseline. The primary outcome measure will be anaerobic threshold. There will also be a subgroup of participants who will undergo muscle biopsy and D2O ingestion to allow an insight into the mechanistic basis behind exercise training response in this age group.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 70 years.
* Sufficient mobility to be able to exercise on a static exercise bike.
* Availability for the entire trial period.
* Sufficient capacity to consent for the trial.

Exclusion Criteria:

* Participants under the age of 70 years.

Participants with a significant past medical history of:

* Myocardial infarction (within last 6 months)
* Unstable Angina
* Heart failure (NYHA class III/IV)
* Uncontrolled Hypertension (BP>160/100)
* Previous stroke/TIA
* Severe respiratory disease inc. known pulmonary hypertension(>25 mmHg), Forced -Expiratory Volume in 1 second <1.5l.
* Brittle asthma / exercise induced asthma
* Known cerebral aneurysm or abdominal aortic aneurysm.
* Cognitive impairment, which may reduce individuals' ability to provide informed consent.
* Inclusion in a recent study which included any form of exercise, taking a drug or ionising radiation.

Exclusion criteria pertaining specifically to muscle biopsies:

* Current use of anticoagulation (i.e. Warfarin/Clopidogrel/Rivaroxaban)
* Any pre-existing clotting disorders known to the patient (i.e. haemophilia).
* Family history of severe bleeding requiring medical intervention.
* Any musculoskeletal deformity or skin conditions making the taking of a biopsy unsuitable as deemed by the medical practitioner taking that sample.
* Lack of capacity to fully consent for the procedure.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09; Primary Completion 2017-10 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Mean anaerobic threshold improvement following 4 week HIT protocol. | 4 weeks
  Measured via cardiopulmonary exercise testing (mls/kg/min and absolute value L/kg). Pre-Post testing.

SECONDARY OUTCOMES:
Mean VO2 peak improvement following 4 week HIT protocol. | 4 weeks
  Measured via cardiopulmonary exercise testing (mls/kg/min and absolute value L/kg). Pre-Post testing.
Muscle protein synthesis | 4 weeks
  Assessment of D2O evaluated muscle protein synthesis following HIT programme. Using mass spectrometry for analysis of stable isotope uptake during training program (arbitrary units).
Body composition | 4 weeks
  DXA changes in body composition (lean muscle mass (%), fat mass (%) and bone density g/cm3)) following a HIT programme
Muscle architecture | 4 weeks
  Ultrasound scans used to assess changes in lean muscle mass and architecture following a HIT programme (mm and % pennation angle change).
Feasibility | 4 Weeks
  Determination of frail elderly patient adherence to HIT programme (number of scheduled sessions successfully completed within 28 days).
Quality of life improvement | 4 weeks
  Quality of life questionnaires to measure subjective outcomes (EQ-5D questionnaire)
Daily Activity Level | 4 weeks
  Activity questionnaire to quantify habitual physical activity (IPAQ questionnaire)
Physical Activity Score | 4 weeks
  Subjective assessment of physical ability (DASI questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: John Williams, BSc MBChB FRCA PhD, Principal Investigator — Nottingham University
Locations (1):
- School of Graduate Entry Medicine, Royal Derby Hospital, Derby, Derbyshire, United Kingdom